CLINICAL TRIAL: NCT07060235
Title: Lumbal Disk Hernili Hastalarda Fasyal Egzersiz Tabanlı Mobil Uygulama Geliştirilmesi ve Etkinliğinin Araştırılması
Brief Title: Development of a Fascial Training Based Mobile Application and Investigation of Its Effectiveness in Patients With Disc Herniation
Acronym: Fascia-M
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BaskentU-FTR-FA-02
Record Dates: First submitted 2025-02-06; First posted 2025-07-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Disease; Lumbal Disc Herniation
Keywords: fascia; mobile app; disc herniation
MeSH Terms: conditions — Intervertebral disc disease; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fascial exercise (Active Comparator): Fascial exercises are a systematic set of movements and manual techniques that target the fascia-the body's connective tissue network-with the aim of improving or maintaining its elasticity, hydration, mobility, and functional integrity. These exercises seek to enhance gliding between fascial layers, reduce tissue restrictions, improve neuromuscular coordination, and alleviate chronic musculoskeletal pain.Fascia is not merely a passive structure; it functions as an active sensory organ containing proprioceptors, nociceptors, and mechanoreceptors.
  This exercise system will first be taught to the patient by a physiotherapist, then a home brochure will be given and the patient will be given 14 days to practice it at home.
  Interventions: Other: fascial exercise home brochure
- Fascial exercise based mobile application (Active Comparator): Individuals in this arm will do fascia exercises at home through a mobile application as home exercises. These exercises would be taught to the participant by the physiotherapist in the clinical setting and then the participant would be allowed to install a mobile application on their phone. The name of this mobile application is Fascia-M. This mobile application will be developed by the researcher of this study during the study process.
  Interventions: Other: Fascial exercise based mobile application
- lumbal stabilization (Active Comparator): Within the scope of this study, lumbar stabilization exercises will be applied to a specific group of participants within a home-based exercise program. The program is structured to support individuals' activities of daily living, maintain spinal health and improve muscle balance in the lumbar region. Lumbar stabilization exercises consist of controlled movements that target the deep spinal stabilizer muscles (especially m. transversus abdominis and m. multifidus) and contribute to maintaining the spine in a neutral position.
  Interventions: Other: lumbal stabilizasyon home brochure

INTERVENTIONS:
Other: fascial exercise home brochure — Fascia exercises are taught by the physiotherapist in the clinical setting and if the exercises are performed incorrectly, intervention is made and the correct exercise is taught. At home, the individual is motivated and monitored with an exercise diary. He/she remembers the exercises from the home brochure.
  Arms: Fascial exercise
Other: Fascial exercise based mobile application — Fascia exercises are taught by the physiotherapist in the clinical setting and if the exercises are performed incorrectly, intervention is made and the correct exercise is taught. At home, the individual is motivated and monitored with an exercise diary. Performs the exercises by watching videos on the mobile application. The physiotherapist intervenes in motivation with instant notifications via the mobile application.
  Arms: Fascial exercise based mobile application
Other: lumbal stabilizasyon home brochure — Participants assigned to the intervention group will receive a structured home-based lumbar stabilization exercise program designed to improve spinal stability, core muscle control, and functional performance. The program will target deep trunk stabilizer muscles, including the transversus abdominis and multifidus, through low-load, motor control-based exercises.
  The intervention will last for 14 days, with exercises to be performed 3 times for everyday, Each session will last approximately 20-30 minutes and consist of:
  Warm-up (1 minutes): Breathing exercises and gentle mobility
  Core Stabilization (15-20 minutes): Exercises such as abdominal hollowing, bridging, bird-dog, side plank, and dead bug - progressing from static holds to dynamic movements as tolerated
  Cool-down (1 minutes): Light stretching and relaxation
  Arms: lumbal stabilization

SUMMARY:
This study will compare three different groups for lumbar disc herniation. The first group will do fascia exercises via a mobile application, the second group will do fascia exercises via a home leaflet, and the third group will do lumbar stabilization exercises via a home leaflet. Since there is not yet a mobile application that includes fascia exercises, this application will be made available to patients for home use after it is developed during the study.

The physiotherapist will teach the exercises in the clinical setting in three different groups.

DETAILED DESCRIPTION:
In the study, 20 people in three different groups with a drop-out rate of twenty percent will participate in the study. This number is 60 people in total.

In the study, fascia exercises will be applied at home with the mobile application named Fascia-M for the first group, fascia exercises will be applied at home with the home brochure for the second group, and lumbar stabilization exercises will be applied at home with the home brochure for the third group. Visual pain scale, Tampa kinesiophobia scale, SF-12 Quality of Life Questionnaire, Pittsburg Sleep Quality Scale, modified schober test, digital inclinometer measurements will be applied and evaluated by the physiotherapist before and after the study.

ELIGIBILITY:
Exclusion Criteria:

* Mobile on Android devices have the competence to use the application
* No neurological deficit
* painkillers during the treatment process
* They are volunteer individuals who do not use medication

İnclusion Criteria:

* speak Turkish, and have Turkish literacy.
* included lumbar
* diagnosed with disc herniation with doctor's diagnosis
* participants is between the ages of 20-55,
* able to use mobile technology
* willing to participate in the study individuals with

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Development of a Fascial Exercise Based Mobile Application and Investigation of Its Effectiveness in Patients with Disc Herniation | 14 days after the start of the exercise programme
  Change in self-reported low back pain intensity as measured by the Visual Analog Scale (VAS). The VAS is a unidimensional pain assessment tool consisting of a 10 cm horizontal line anchored by "no pain" (0 cm) and "worst imaginable pain" (10 cm). Participants will mark their current pain level on the line. The distance (in cm) from the left end to the mark will be recorded as the pain score.

SECONDARY OUTCOMES:
Development of a Fascial Exercise Based Mobile Application and Investigation of Its Effectiveness in Patients with Disc Herniation | 14 days after the start of exercise programme
  Change in lumbar functional disability assessed using the Oswestry Disability Index (ODI). The ODI consists of 10 sections measuring the degree of disability in daily living activities due to low back pain. Total scores range from 0% (no disability) to 100% (maximum disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent Universty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: fascial fıtness — https://www.anatomytrains.com/fascialfitness/fascial_fitness1.pdf
- Available data/document: statics: fascial tarining — https://www.anatomytrains.com/fascialfitness/fascial_fitness1.pdf — fascia and mobile app